CLINICAL TRIAL: NCT06033339
Title: Etude du rôle Des microARNs Dans la Physiopathologie de la fièvre méditerranéenne Familiale
Brief Title: Assessment of microRNAs Role in Familial Mediterranean Fever FMF Pathophysiology
Acronym: miRinFMF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0296 - UF 8310
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Familial Mediterranean Fever
Keywords: MEditerranean FeVer MEFV gene; micro ribonucleic acid miRNA
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Among the 40 subjects to be enrolled: 10 are MEFV homozygous patients, 10 are symptomatic MEFV heterozygous patients, 10 are asymptomatic MEFV heterozygous patients and 10 are control subjects. All enrolled patients receive the same intervention (biological sample collection).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood Sampling (Other): Collection of 10 ml of blood on EDTA tube during:
  * Standard check-up visit as a part of the standard monitoring of the disorder for homozygous and symptomatic heterozygous patients
  * Specific study visit for asymptomatic heterozygous patients
  * Presurgery blood test for control subjects
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Collection of 10 ml of blood on EDTA tubes per patient. Once collected, the blood tubes will be transported within 24 hours to the IRB (Biotherapy Research Institute) of Montpellier University Hospital, where the monocytes will be isolated by magnetic sorting on the basis of expression of surface marker CD14+, after a preliminary step of Ficoll. Monocytes will then be frozen in nitrogen at -196°C until use (biobank).Gain-of-function experiments will then be performed on monocytes by transfecting them with the microRNA of interest or control. The expression of the pyrin protein and its phosphorylation rate will be evaluated after induction by immunoprecipitation experiments followed by western blot. The activity of the pyrin inflammasome will also be studied by looking at pyroptosis and toxicity rate using LDH test. All these experiments will be carried out in the absence and in the presence of the microRNA in order to study its role in the pathophysiology of FMF.

SUMMARY:
Familial Mediterranean Fever (FMF) genetic diagnosis is well established for homozygous patients. On the other hand, although heterozygous individuals are theoretically healthy carriers, 1/3 of them will develop clinical symptoms of FMF and could benefit from prophylactic treatment. This suggests that the disorder expression mechanisms are not fully elucidated to date. The preliminary results obtained at the Institute for Regenerative Medicine and Biotherapy (IRMB) suggest the involvement of an epigenetic mechanism in FMF pathogenesis, and our laboratory has strong arguments as to the involvement of microRNAs (in particular miR-326) which are negative regulators of gene expression.

This study is exploratory and aims to validate the role of miRNAs in the clinical expression of FMF in patients, thus to explore the epigenetic mechanisms that may explain the variability of expression of this disorder.

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF) is a rare autoinflammatory disorder due to mutations in the MEFV (MEditerranean FeVer) gene, that causes recurrent episodes of fever and acute serositis (peritoneum, pleura, synovium) beginning in early childhood.

MEFV gene identification allowed the development of a genomic sequencing test to confirm the diagnosis. The most frequent mutations are M680I, M694V, V726A and M694I, located in exon 10. This gene encodes the protein pyrin, which, following a pro-inflammatory stimulus, is capable of assembling a multi-protein complex to form the pyrin inflammasome. MEFV gene mutations lead to an alteration of its expression in innate immune system cells in FMF patients, causing a dysregulation of the immune response, which results in the abnormal secretion of certain proinflammatory cytokines such as IL-1β and IL-18.

FMF is an autosomal recessive disorder. Thus, heterozygous individuals are theoretically healthy carriers. Nevertheless, in nearly 1/3 of patients with clinical symptoms of FMF, a single heterozygous mutation is found. To date, there is no biological marker to distinguish heterozygous individuals who will develop the disease from those who remain healthy carriers, hence diagnostic errors and delays in treatment. Several hypotheses have been put forward to explain this variation in mutation expression, whether it is the environment, the involvement of other genes, or the involvement of epigenetic modifiers.

Among the mechanisms that regulate gene expression, microRNAs (miRNAs),which are small non-coding RNAs, negatively regulate gene expression at the post-transcriptional level by binding to sequences located mainly in the region 3'UTR of gene mRNA. Many publications report that they are abnormally expressed in various pathologies. Very recently, this has been reported for FMF. Several studies have focused on miRNAs as biomarkers of FMF, without evaluating their role in FMF pathogenesis.

Assessing the role of miRNAs specifically targeting the MEFV gene in myeloid cells (especially monocytes), and the functional impact of their modulation in these cells, would deepen our understanding of FMF physiopathology. If a miRNA specifically targeting MEFV has a proven role in FMF pathophysiology, it could ultimately prove to be a prognostic biomarker of the disorder for heterozygous patients, or even a future therapeutic target.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥1 year
* Body weight ≥ 10kg
* Homozygous patients group: patients homozygous for MEFV (M694V, M694I, M680I, V726A)
* Symptomatic heterozygous patients group: patients heterozygous for the MEFV gene (M694V, M694I, M680I, V726A) meeting the Yalcinkaya criteria for FMF diagnosis (Fever lasting 6 to 72 hours with at least 3 attacks - Abdominal pain of 6 to 72 hours duration with at least 3 attacks - Chest pain of 6 to 72 hours duration with at least 3 attacks - Arthritis of 6 to 72 hours duration with at least 3 attacks- FMF Family History of FMF)
* Asymptomatic heterozygous patients group: patients heterozygous for the MEFV gene (M694V, M694I, M680I, V726A) who do not meet the Yalcinkaya criteria for FMF diagnosis
* Control subjects group: absence of identified auto-inflammatory disorder

Exclusion Criteria:

* Absence of collection of informed consent of participant or absence of informed consent of the legal representatives/guardians of pediatric participant
* Subjects not registered in Social Security system

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2025-10-02 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
miR-326 expression level quantification | 1 day (at enrollment)
  Analyze the expression levels (quantification) of miRNA miR-326 in blood monocytes within the 4 groups of individuals: homozygous, symptomatic heterozygous, asymptomatic heterozygous for MEFV and control subjects, in order to determine whether or not miR-326 influences the inflammatory response of monocytes.
MEFV expression level quantification | 1 day (at enrollment)
  Analyze the expression levels (quantification) of MEFV gene in blood monocytes within the 4 groups of individuals: homozygous, symptomatic heterozygous, asymptomatic heterozygous for MEFV and control subjects

SECONDARY OUTCOMES:
miR-326 expression level comparison | 1 day (at enrollment)
  Compare the expression levels of miR-326 between symptomatic and asymptomatic heterozygous groups.
MEFV expression level comparison | 1 day (at enrollment)
  Compare the expression levels of MEFV between symptomatic and asymptomatic heterozygous groups.
Blood samples collection | 1 day (at enrollment)
  Create a biobank (freezing monocytes extracted from patient samples) in order to subsequently study other miRNAs
Expression levels of other candidate miRNAs targeting MEFV | 1 day (at enrollment)
  Quantification of the the expression levels of other candidate miRNAs targetting MEFV within the 4 groups of participants. 5 miRNAs will be selected using a methylome study currently being carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Eric JEZIORSKI, MD, Principal Investigator — University Hospital, Montpellier
Locations (4):
- France (4):
  - University Hospital of Nîmes, Nîmes
  - Robert Debré University Hospital of Paris, Paris
  - University Hospital of Paris Kremlin Bicêtre, Paris
  - University Hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No